CLINICAL TRIAL: NCT01522937
Title: A Phase II Study of Individualized Stereotactic Body Radiation Therapy (SBRT) for Intrahepatic Cancer
Brief Title: A Study of Individualized Stereotactic Body Radiation Therapy (SBRT) for Intrahepatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2009-053; HUM00029467 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2011-09-23; First posted 2012-02-01 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Liver Cancer; Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liver cancer patients (Experimental): The aim of this study is to determine the safety and effectiveness of individualized Stereotactic Body Radiation Therapy (SBRT) in patients who either (1) have had previous liver treatments, and/or (2) have primary hepatocellular carcinoma (HCC).
  Interventions: Radiation: individualized Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: individualized Stereotactic Body Radiation Therapy (SBRT) — The individualized SBRT involves two treatment phases. The first phase of treatment involves receiving three fractions of SBRT, followed by a 1-month break and assessment of liver function with a blood test - Indocyanine Green (IC-Green). The second phase of treatment involves receiving two more fractions of SBRT, whose doses are adjusted to account for tolerance of the first phase of treatment.

SUMMARY:
This is a Phase II trial to characterize the safety and efficacy of individualized stereotactic body radiation therapy (SRBT) for patients who have had previous liver treatment or who have primary hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The trial endpoints are toxicity, survival and progression-free survival. DCE-MRI and plasma biomarkers will also be collected to explore their use as tools for treatment individualization in future trials. During the current trial, an indicator of liver function, indocyanine green (ICG), will be used to identify during treatment patients who are at excess risk for radiation-induced liver disease (RILD) so that their radiation dose may be reduced. The model used for individualization will be updated as trial data accrue, so this is an adaptive trial of an individualized therapy. The planned accrual is seventy (70) evaluable patients over three years.

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* life expectancy of at least 12 weeks
* Zubrod performance status of ≤2.
* biopsy proven hepatocellular carcinoma (HCC)
* liver metastases
* a discrete hepatic tumor(s) as defined by the Barcelona46 criteria - for cirrhotic patients, (1) 2 imaging studies showing hypervascular tumor > 2cm, or (2) single imaging study showing hypervascular tumor > 2cm with AFP ≥ 400 ng/mL
* a discrete hypervascular tumor present on two consecutive imaging studies (CT or MRI) with documented growth of > 1cm in diameter
* adequate organ function
* women and men not interested in pregnancy
* must be recovered from the effects of any prior surgery, radiation therapy, chemotherapy and the effects of Radiofrequency Ablation (RFA) or Transcatheter Arterial Chemo Embolization (TACE)
* minimum of 6 weeks following their last surgical procedure, radiation and chemotherapy.

Exclusion Criteria:

* cannot be eligible for a curative liver resection
* uncontrolled ascites clinically evident on physical exam
* known allergy to IC-Green
* known allergy to intravenous iodinated contrast agents
* patients with poor venous access
* patients with metastatic cancer with normal liver function who have not undergone previous liver directed therapy and a single tumor < 6 cm in size.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Cuneo, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Feng M, Suresh K, Schipper MJ, Bazzi L, Ben-Josef E, Matuszak MM, Parikh ND, Welling TH, Normolle D, Ten Haken RK, Lawrence TS. Individualized Adaptive Stereotactic Body Radiotherapy for Liver Tumors in Patients at High Risk for Liver Damage: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Jan 1;4(1):40-47. doi: 10.1001/jamaoncol.2017.2303. PMID 28796864

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liver Cancer Patients
Started | 146
Completed | 146
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 146
Age, Continuous [Mean (Full Range); unit: years] | 65 [25 to 86]
Gender [Count of Participants; unit: Participants]
  Female | 30
  Male | 116

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Local Control at 1 Year Post Treatment
Description: For this study, local control is defined as the lack of progressive local disease following CR (Complete Response) or PR (Partial Response), or lack of progressive local disease in patients with non-evaluable disease, who have no progressive elevation in serum tumor markers.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 102
percentage of patients | 99 [97 to 100]

2. Secondary Outcome: The Percentage of Patients Alive Without Progression at 1 Year
Description: Progression is defined as a greater than or equal to 20% growth of a lesion from the smallest lesion measurement
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 102
percentage of patients | 62 [53 to 71]

3. Secondary Outcome: The Percentage of Patients Alive at 1 Year
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 102
percentage of patients | 67 [58 to 78]

4. Secondary Outcome: The Number of Patients Who Experience Grade 4+ Hepatotoxicity
Description: Grade 4 toxicities are life threatening toxicities that require urgent attention.
Time Frame: 1 Year
Measure: Number; unit: patients
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 102
patients | 0

5. Secondary Outcome: The Number of Patients That Experience Grade 4+ Gastrointestinal Bleeding
Description: Grade 4 toxicities are life threatening toxicities that require urgent attention.
Time Frame: 1 Year
Measure: Number; unit: patients
Arm/Group | Liver Cancer Patients
Number analyzed (Participants) | 102
patients | 0

ADVERSE EVENTS:
Arm/Group | Liver Cancer Patients
Serious Adverse Events (participants affected / at risk) | 22/146
Other Adverse Events (participants affected / at risk) | 81/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liver Cancer Patients (N=146)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Social circumstances - Other (Social circumstances) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Psychiatric disorders - Other (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (3)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liver Cancer Patients (N=146)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 21 (22)
Oral pain (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 5 (6)
General disorders and administration site conditions - Other (General disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 33 (38)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 21 (24)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 12 (18)
Serum amylase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 7 (12)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 3 (3)
Personality change (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (10)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (11)
Chills (General disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 6 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8)
Fatigue (General disorders) | 64 (94)
Fever (General disorders) | 1 (2)
Psychiatric disorders - Other (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes